CLINICAL TRIAL: NCT02773173
Title: Individualized Pneumoperitoneum Pressure in Colorectal Laparoscopic Surgery Versus Standard Therapy (IPPCollapse II)
Brief Title: Individualized Pneumoperitoneum Pressure in Colorectal Laparoscopic Surgery Versus Standard Therapy (IPPCollapse-II)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto de Investigacion Sanitaria La Fe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IPPCollapse-II
Record Dates: First submitted 2016-05-02; First posted 2016-05-16 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Surgery; Laparoscopy
Keywords: Colorectal Laparoscopic Surgery
MeSH Terms: interventions — indolepropanol phosphate; signal peptide peptidase

STUDY DESIGN:
Intervention Model Description: neuromuscular blocking agents as type of drug
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Pneumoperitoneum Pressure (Experimental): In Individualized Pneumoperitoneum Pressure (IPP) group, measures to optimize and individualize intra-abdominal pressure (PIA) will be apply.
  Interventions: Procedure: IPP in colorectal laparoscopic surgery
- Standard Pneumoperitoneum Pressure (Other): In Standard Pneumoperitoneum Pressure (SPP) group, a conventional operation without optimization measures and PIA preset to 12 mmHg will be conducted.
  Interventions: Procedure: SPP in colorectal laparoscopic surgery

INTERVENTIONS:
Procedure: IPP in colorectal laparoscopic surgery — Deep neuromuscular blockade can only be reversed with sugammadex, so in the IPP group, it will be used as neuromuscular blocking agent and its effect will be reversed with sugammadex (4mg / kg) at the end of the surgery. During surgery: deep neuromuscular blockade (PTC 1-5), Protective ventilation strategy, Optimal position and Pre stretching as a tool to decrease intraabdominal pressure maintaining optimal workspace.
  Arms: Individualized Pneumoperitoneum Pressure
Procedure: SPP in colorectal laparoscopic surgery — A depolarizing neuromuscular blocking will be used (as routine clinical practice at each center) to maintain moderate neuromuscular blockade and its effect will be reversed with anticholinesterase at the end of the surgery. During surgery: Moderate neuromuscular blockade ( TOF 2-4) , position to surgeon criteria, no prestretching and Protective ventilation. Fixed IAP (12mmHg).
  Arms: Standard Pneumoperitoneum Pressure

SUMMARY:
The purpose of this study is to assess the post-operative recovery quality of the Individualized Pneumoperitoneum Pressure Therapy in Colorectal laparoscopic surgery versus standard therapy using a quality validated scale of postoperative recovery of their stay in the Post-Anaesthesia Recovery Unit.

DETAILED DESCRIPTION:
In the last two decades laparoscopic surgery has settled as a less invasive surgical approach compared to open surgery. It is associated with lower perioperative morbidity and hospital stay. There is growing evidence that increased intra-abdominal pressure (IAP), even for short periods of time, is associated with increased perioperative morbidity (pain, increased inflammatory markers peritoneal injury worse splanchnic perfusion abnormalities hemodynamic and ventilatory ...).

The study is a prospective multicenter randomized clinical intervention trial to assess the impact of IAP individualization strategy (IPP-Individualized pneumoperitoneum Pressure) relative to a IAP standard strategy (SPP-Standard pneumoperitoneum Pressure) using a validated scale (VAS) (PQRS- Postoperative Quality of Recovery Scale). Postoperative pain in the first 24 hours (area under VAS curve , opioid rescue, referred pain to the shoulder) and surgical stress and inflammatory markers (neutrophil/lymphocyte, ratio,C-reactive protein, interleukin-6, procalcitonin) are also measured. Postoperative complications are evaluated by Clavier-Dindo classification.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Classification of the American Society of Anesthesiologists (ASA I-III)
* No cognitive deficits
* Signed informed consent prior to surgery

Exclusion Criteria:

* Emergency surgery
* Pregnancy or lactation
* Immune disorders
* Kidney or liver disease or advanced-stage cardiopulmonary
* Patient refusal to participate in the study
* Patients under 18 years or inability to consent
* Associated neuromuscular disorders, contraindication for the use of rocuronium/ sugammadex, allergy or hypersensitivity to rocuronium / sugammadex

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Change in Postoperative Quality of Recovery Scale (PQRS) Physiologic Domain | Up to postoperative day 3. This is a longitudinal outcome.
  The primary outcome of the IPPCollapse II study is the recovery of the Physiologic' component of the PQRS score over the assessed time points. The PQRS is a validated multidimensional patient Reported Outcome (PRO) tool designed to assess patients' recovery to baseline status in the postoperative period (www.postopqrs.com). In every patient a baseline measurement of PQRS is performed prior to surgery. After surgery, the measurement of the PQRS is repeated at 15 min (T15) and at 40 min (T40) after arrival in the PACU, as well as in the ward on the morning of postoperative day ( POD) one and three. Physiologic domain includes 9 variables scored from 1-3, 9 is the minimum and worse recover and 27 is the maximum and full recover. But recovery is related to baseline. Each patient is scored at the predefined time points and is classified as either 'recovered' if the score reaches at least the predetermined baseline score or 'not recovered' .

SECONDARY OUTCOMES:
Chnge Postoperative Quality of Recovery Scale (PQRS) | Up to postoperative day 3. This is a longitudinal outcome.
  The PQRS domains, 'nociceptive', 'emotional', 'cognitive', and 'functional' components, as well as the 'overall score' are used as secondary outcomes. In every patient a baseline measurement of PQRS is performed prior to surgery. After surgery, the measurement of the PQRS is repeated at 15 min (T15) and at 40 min (T40) after arrival in the PACU, as well as in the ward on the morning of postoperative day ( POD) one and three. Nociceptive and emotional domains are scored from 1-5 ( from worse to better) and include 4 variables. Functional domain is scored from 1-3 ( From worse to better) and include 4 variables, and cognitive is depicted as recover or not versus baseline score.
Daily postoperative complications until hospital discharge (Clavien-Dindo) | Up to postoperative day 28
  Postoperative complications clavien dindo classification
Basic features of airway pressures (plateauP, peakP, pulmonary Compliance) | Up to 300 minutes during surgical intervention
  Airway pressures in cmH2O
Intraabdominal pressure | Up to 300 minutes during surgical intervention
  Intraabdominal pressures in mm Hg
Intraabdominal volume | Up to 300 minutes during surgical intervention
  Intraabdominal pressures in ml
Spontaneous / coughing movements . | Up to 300 minutes during surgical intervention
  yes or no
Substudy- Hepatic perfusion during pneumoperitoneum.Plasma disappearance rate of indocyanine green (PDRICG) | Up to 300 minutes during surgical intervention
  Plasma disappearance rate of indocyanine green
Change in Surgical stress and inflammatory markers | Up to postoperative day 3. This is a longitudinal outcome
  (neutrophil/lymphocyte ratio, C-reactive protein,interleukin-6 and procalcitonin).

CONTACTS AND LOCATIONS:
Overall Officials: Óscar Díaz, Principal Investigator — Instituto de Investigación Sanitaria La Fe
Locations (1):
- Hospital universitario y Politécnico La Fe, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diaz-Cambronero O, Mazzinari G, Flor Lorente B, Garcia Gregorio N, Robles-Hernandez D, Olmedilla Arnal LE, Martin de Pablos A, Schultz MJ, Errando CL, Argente Navarro MP; IPPColLapSe II study investigators. Effect of an individualized versus standard pneumoperitoneum pressure strategy on postoperative recovery: a randomized clinical trial in laparoscopic colorectal surgery. Br J Surg. 2020 Nov;107(12):1605-1614. doi: 10.1002/bjs.11736. Epub 2020 Jun 7. PMID 32506481
- [Derived] Diaz-Cambronero O, Mazzinari G, Errando CL, Schultz MJ, Flor Lorente B, Garcia-Gregorio N, Vila Montanes M, Robles-Hernandez D, Olmedilla Arnal LE, Martin-De-Pablos A, Marques Mari A, Argente Navarro MP; IPPCollapse-II study group. An individualised versus a conventional pneumoperitoneum pressure strategy during colorectal laparoscopic surgery: rationale and study protocol for a multicentre randomised clinical study. Trials. 2019 Apr 3;20(1):190. doi: 10.1186/s13063-019-3255-1. Erratum In: Trials. 2020 Jan 13;21(1):70. doi: 10.1186/s13063-020-4055-3. PMID 30944044